CLINICAL TRIAL: NCT01892865
Title: Use of Predictive Modeling to Improve Operating Room Scheduling Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IIR 12-113
Record Dates: First submitted 2013-07-01; First posted 2013-07-08 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-05

CONDITIONS: Operating Room Scheduling
Keywords: Operating room utilization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Historical means method (Active Comparator): Operative time will be predicted using historical service means. Schedule will be constructed using this time
  Interventions: Other: Scheduling using historical means
- Predictive Modeling System (PMS) (Experimental): Operative time will be predicted using a regression model. Schedule will be constructed using this time
  Interventions: Other: Scheduling using regression modeling system

INTERVENTIONS:
Other: Scheduling using historical means — Scheduling will be performed taking into account historical means only for anesthetic, operative, and turn around time
  Arms: Historical means method
Other: Scheduling using regression modeling system — A regression model that uses predictor of operative length will be used to predict operative, anesthetic, and turn around time length
  Arms: Predictive Modeling System (PMS)

SUMMARY:
This study compares two different methodologies of scheduling cases in the operating room.

DETAILED DESCRIPTION:
The goal of the proposed study is to address the efficacy of a scheduling methodology that uses a regression-based predictive modeling system (PMS) to calculate operative and anesthetic time length. The investigators hypothesize that compared to the traditional scheduling system (TSS) that calculate operative length using historic means, case allocation in an operating room using the PMS will improve scheduling precision, increase operative volume and increase Operative Suite (OS) personnel satisfaction, without having adverse impact on patient outcomes. The investigators will evaluate this hypothesis using a randomized block design in two operating rooms of a single surgical specialty for a total of 100 operative days per arm.

ELIGIBILITY:
Inclusion Criteria:

* The only requirement for including a day in the study will be that all the procedures performed in that specific day have been previously performed in our hospital at least 5 times a year for each of the last three years. This rule will encompass the vast majority of the performed vascular procedures in our facility. Setting the threshold at a minimum of 5 cases per year is essential to assure that some data will be available to calculate the expected length of the case with either the traditional or the predictive modeling system. If a case is performed in a day when the scheduling imprecision is supposed to be calculated using the PMS but modeling data do not exist, then the anticipated length of this case will be calculated using the historic means.
* Surgery cancellation after the first case will not disqualify that day from inclusion in the study. If the cancellation occurs in the last case of the sequence for the specific day then no particular intervention will be taken. The anticipated end of the surgical day will reset to the end of the last case that took place, and all the imprecision calculations will be performed as described below. If the cancellation occurs in one of the intermediate cases, then the end of the operative day will reset to reflect the removal of the cancelled case.

Exclusion Criteria:

A day will be excluded from the study when any of the following occur (based on historical data the investigators anticipate 10-15% of the operative days to meet the exclusion criteria):

* Only one or no cases have been scheduled for the entire operative day
* An emergency case is added as first case, or in between the scheduled cases.
* The operative day falls during a major holiday week (Thanksgiving, Christmas, New Year). The schedule during these time periods tends to be fragmented, cancellation rates are high, and cases are frequently performed with back-up teams only. All these factors may distort the findings.
* There is an unusual case in the schedule that does not meet the minimum requirement of 5 previous operations on a yearly basis for the last three years.
* The first case of the day is cancelled

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 735 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Kougias, MD MSc, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX; David H. Berger, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kougias P, Tiwari V, Sharath SE, Garcia A, Pathak A, Chen M, Ramsey D, Barshes NR, Berger DH. A Statistical Model-driven Surgical Case Scheduling System Improves Multiple Measures of Operative Suite Efficiency: Findings From a Single-center, Randomized Controlled Trial. Ann Surg. 2019 Dec;270(6):1000-1004. doi: 10.1097/SLA.0000000000002763. PMID 29697450

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Calendar days during which vascular surgery operations were performed were randomly scheduled using either the Historical Means or the Predictive Modeling System methodologies. Please, note that unit of randomization was operative days, not patients
Pre-assignment Details: Operative days that were on holidays, or when staff surgeons were out of town were excluded. Similarly, did not schedule any cases during the re-calibration of the predictive models
Units Other Than Participants: Operative Days
Period: Overall Study
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Started | 356; 107 Operative Days (107 operative days scheduled with the Historical Means method were included) | 379; 100 Operative Days (100 operative days scheduled with the Predictive Modeling System method were included)
Completed | 356; 107 Operative Days | 379; 100 Operative Days
Not Completed | 0; 0 Operative Days | 0; 0 Operative Days

BASELINE CHARACTERISTICS:
Units Other Than Participants: Operative Days
Groups:
- Total: Total of all reporting groups
Arm/Group | Historical Means Method | Predictive Modeling System (PMS) | Total
Number analyzed (Participants) | 356 | 379 | 735
Number analyzed (Operative Days) | 107 | 100 | 207
Age, Customized [Mean (Standard Deviation); unit: Years] | 62 (8) | 62.5 (10) | 62.5 (10)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Males | 351 | 373 | 724
  Sex: Females | 5 | 6 | 11
Available operative days for randomization [Count of Units; unit: Operative Days] | 107 | 100 | 207

OUTCOME MEASURES:

1. Primary Outcome: Difference Between the Actual and Predicted Length of Operative Day (in Minutes)
Description: The scheduling imprecision between the two scheduling approaches will be compared. Scheduling imprecision is defined as the difference between the actual and predicted length of operative day.
Time Frame: Three years
Population: We analyzed data from 107 operative days in the HM arm, and 100 days in the PMS arm
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Number analyzed (Participants) | 107 | 100
Minutes | 30.8 (99) | 7.2 (67)
Statistical Analysis 1: Comparison: Historical Means Method vs Predictive Modeling System (PMS); The null hypothesis was that there would be no difference in predictive imprecision for the end of the operative day between the two arms; Test type: Superiority or Other; p = 0.024, t-test, 2 sided; Mean Difference (Net) = 23.6, 95% CI 2-sided [3.15 to 44]
Statistical Analysis 2: Comparison: Historical Means Method vs Predictive Modeling System (PMS); Null hypothesis: There would be no difference in throughput between the two arms; Test type: Superiority or Other; p = 0.04, Poisson regression; Risk Ratio (RR) = 1.16, 95% CI 2-sided [1.01 to 1.34]

2. Secondary Outcome: Difference in Throughput
Description: Difference in total number of cases scheduled per unit of time analyzed between the two study arms
Time Frame: Three years
Population: Operative days
Measure: Number; unit: Operations/day analyzed
Units Other Than Participants: Operative Days
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Number analyzed (Participants) | 356 | 379
Number analyzed (Operative Days) | 107 | 100
Operations/day analyzed | 3.33 | 3.79
Statistical Analysis 1: Comparison: Historical Means Method vs Predictive Modeling System (PMS); Null hypothesis was that there was no difference in throughput between the two scheduling methods; Test type: Superiority or Other; p = 0.04, Poisson Regression; Risk Ratio (RR) = 1.16, 95% CI 2-sided [1.01 to 1.34]

3. Secondary Outcome: Operative Suite Personnel Job Satisfaction
Description: Comparison of job satisfaction between study arms using three domains of the Maslach Burnout Inventory: Depersonalization (range 0-17, score of 17 indicates worse depersonalization). Emotional Exhaustion (range: 0-36, score of 36 is the worse). Personal accomplishment (range 1-60, score of 60 is best).
Time Frame: Three years
Population: Health care providers
Measure: Mean (Full Range); unit: units on a scale
Units Other Than Participants: Responses
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Number analyzed (Participants) | 21 | 21
Number analyzed (Responses) | 61 | 53
units on a scale
  Depersonalization | 3.23 [0 to 17] | 2.04 [0 to 10]
  Emotional Exhaustion | 11.82 [0 to 29] | 10.03 [0 to 36]
  Personal Accomplishment | 37.51 [15 to 48] | 40.47 [21 to 48]
Statistical Analysis 1: Comparison: Historical Means Method vs Predictive Modeling System (PMS); Null hypothesis: There would be no difference in personnel satisfaction between the groups; Test type: Superiority or Other; p = 0.04, t-test, 2 sided

4. Secondary Outcome: Complications: A Composite Endpoint of Death, Myocardial Infarction, Bleeding, Amputation
Description: Comparison of the perioperative (30-day postoperative) composite endpoint of death, myocardial infarction, bleeding, amputation between the two study groups
Time Frame: Three years
Population: Patients
Measure: Count of Participants; unit: Participants
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Number analyzed (Participants) | 356 | 379
Participants | 8 | 12
Statistical Analysis 1: Comparison: Historical Means Method vs Predictive Modeling System (PMS); Null hypothesis was that there would be no difference in the adverse event rates between the two scheduling methodologies; Test type: Superiority or Other; p = 0.44, Chi-squared

ADVERSE EVENTS:
Time Frame: Randomization unit in this study was operative days; thus, no adverse events were expected.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Historical Means Method | Predictive Modeling System (PMS)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No